CLINICAL TRIAL: NCT03704896
Title: PRospective Observational Multicentre Study on VAriability of Lung Function in Stable PCD Patients
Acronym: PROVALF-PCD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southampton (Other)
Collaborators: University of Bern (Other); Assistance Publique - Hôpitaux de Paris (Other); University of Melbourne (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital, Motol (Other); Copenhagen University Hospital, Denmark (Other); University Hospital Muenster (Other); Hacettepe University (Other); University of Cyprus (Other); University of Sydney (Other); Ruhr University of Bochum (Other); Marmara University (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Meyer Children's Hospital IRCCS (Other); Federico II University (Other); Bambino Gesù Hospital and Research Institute (Other); University of Valencia (Other); Universidade Nova de Lisboa (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: PROVALF
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lung function measurement — Spirometry-derived lung function measurements

SUMMARY:
Using routinely collected clinical data, this study aims to quantify intra-individual (i.e. in the same individual) variations between measurements of lung function in stable patients with primary ciliary dyskinesia (PCD), a rare genetic disease that causes lung damage.

DETAILED DESCRIPTION:
Background

Lung function measurements are commonly used in PCD to monitor disease progression. Spirometry measurements are taken every 3 months and results are compared to established references, adjusted for age, height and ethnicity. Results are also compared to previous measurements from the same patient at earlier appointments. However, little is understood of the impact of intra-individual variability and the extent of spontaneous variations in these comparisons.

One of the priorities for respiratory research in the UK is to understand factors involved in determining different outcomes for lung function.[1] The precision of measurements done on the same individual conducted by different people, in different settings and using different equipment is not entirely known. Importantly, previous studies in healthy children assessing intra-individual variability have shown variations of up to 1.2 z-scores in spirometry parameters over the course of 1 year.[2] Within test-variability and daily repeatability can range from 2 to10% FEV% predicted in young healthy children.[3],[4]

In PCD, deterioration of lung function does not follow a pre-defined pattern.[5] However, none of the published studies on lung function in PCD to date have taken into consideration the imprecision of individual and repeated measurements on the same individual over time. Personal experience and unpublished small retrospective assessments suggest that there is considerable variability.

Key research question

Quantify intra-individual (i.e. in the same individual) variations between measurements of lung function in stable patients with primary ciliary dyskinesia (PCD), a rare genetic disease that causes lung damage.

Study design

Prospective multicentre cohort study using routinely collected clinical data to evaluate natural variability of lung function measurements in stable PCD patients.

The primary end-point is to assess intra-individual variations between repeated measures of lung function parameters. Secondary end-points include: a) Inter-individual variations between repeated measures of lung function parameters and correlations with baseline measures; b) intra- and inter-individual variation between repeated measures of lung function parameters during exacerbation.

Participants will be approached by their clinicians and asked to sign a consent form to allow for their anonymised routinely collected clinical data to be entered into the study. Routine clinical data will be collected at PCD follow-up clinics in participating centres. These data are already collected for clinical purposes and will be anonymised locally. Non-identifiable data will be entered into the study database by a member of the clinical team of the participating centre. The study coordinating centre (University of Southampton) will only have access to the anonymised dataset.

The data collection period will last 18 months (6 months for patients recruitment and 12 months for patient follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Children (>5 years of age) and adults being follow-up for PCD
* Availability of at least minimal dataset (spirometry data), at least every 6 months
* Outpatients and/or in-patients

Exclusion Criteria:

* Children < 5 years of age
* Regular interval between spirometry testing > 6 months

Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with PCD under regular follow-up at one of the centres participating in the study.
Sampling Method: Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Intra-individual variability of FEV1 z-scores | up to one-year follow-up period
  Natural intra-individual variability of FEV1 z-score in patients that are not experiencing an episode of chest exacerbation at the time of lung function measurement.

SECONDARY OUTCOMES:
Inter-individual variability of FEV1 z-scores | up to one-year follow-up period
  Inter-individual variations between repeated measures of lung function parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised centre-specific data will be shared between PROVALF-PCD study and prospective PCD registry and retrospective iPCD cohort, where specifcially requested by centre contributing with data. All parties involved in data transfer will sign an agreement with PROVALF-PCD prior to any data transfer.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Throughout the study, when requested; and at the end of the study, if requested.